CLINICAL TRIAL: NCT03519750
Title: Pharmacokinetics of Intravenous, Rectal, Intravesical, Vaginal, and Transdermal Administration of Exogenous Melatonin in Healthy Female Volunteers: a Crossover Study
Brief Title: Pharmacokinetics of Intravenous, Rectal, Intravesical, Vaginal, and Transdermal Melatonin in Healthy Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dennis Bregner Zetner (Other)
Collaborators: Copenhagen University Hospital, Denmark (Other); RepoCeuticals ApS (Unknown); Herlev Hospital (Other)
Responsible Party: Sponsor-Investigator, Dennis Bregner Zetner, Principal Investigator, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-000997-13
Record Dates: First submitted 2018-04-16; First posted 2018-05-09 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Melatonin; Pharmacokinetics; Safety
Keywords: Melatonin; Safety; Pharmacokinetics
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Each volunteer will have melatonin administered through all five routes of administration, and will have a wash-out of a minimum of 7 days between each administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Intravenous melatonin (Active Comparator): Intravenous administration, making it possible to calculate bioavailability for other routes of administration
  Interventions: Drug: Melatonin 25 mg
- Rectal melatonin (Experimental): Rectal administration of melatonin
  Interventions: Drug: Melatonin 25 mg
- Intravesical melatonin (Experimental): Intravesical administration of melatonin
  Interventions: Drug: Melatonin 25 mg
- Vaginal melatonin (Experimental): Vaginal administration of melatonin
  Interventions: Drug: Melatonin 25 mg
- Transdermal melatonin (Experimental): Transdermal administration of melatonin
  Interventions: Drug: Melatonin 25 mg

INTERVENTIONS:
Drug: Melatonin 25 mg — 24-48 hour monitoring of plasma melatonin as well as adverse events.

SUMMARY:
We will investigate the safety and pharmacokinetics of melatonin, when administered rectally, intravesically, vaginally and transdermally. We will recruit 10 healthy female volunteers. The volunteers will have melatonin administered over 5 days; intravenously, rectally, intravesically, vaginally and transdermally. The participants will be followed for 24-48 hours with blood samples and questions about adverse events. There will be a wash-out between each session of a minimum of 7 days.

ELIGIBILITY:
Inclusion criteria:

* Healthy female
* 20-40 years old
* BMI 18-30

Exclusion criteria:

* Inability to understand Danish, written or spoken.
* Current use of melatonin or other hypnotics/sedatives
* Current pregnancy (a positive urine-HCG; the subjects will be tested prior to each study session)
* Breast feeding
* Current alcohol or drug abuse (defined as over 5 units of alcohol per day, or any usage of illegal drugs)
* Mental illness (defined as being in medical treatment)
* Serious comorbidity (American Society of Anesthesiologists (ASA) physical status 3-4)
* Participation in other clinical trials less than 1 month prior to current study
* Night-shift work within the last 14 days prior to study
* Planned night-shift work within the study period
* Known and diagnosed sleep-disorder (defined as being in current medical treatment)
* Plasma hemoglobin <7.8 mmol/L (measured when screening participants)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — They need to be female, in order to receive vaginal administration of melatonin
Enrollment: 10 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of melatonin | Baseline, 0 minutes, 10 minutes, 20 minutes, 30 minutes, 40 minutes, 50 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 24 hours
  Plasma concentration of melatonin
Plasma concentration of melatonin | Baseline, 0 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 16 hours, 24 hours, 48 hours
  Plasma concentration of melatonin

SECONDARY OUTCOMES:
Karolinska Sleepiness Scale | 0 minutes, once hourly for 8 hours, and again at 24 hours
  Scale which evaluates tiredness of participants
Simple Reaction Time Test | 0 minutes, once hourly for 8 hours, and again at 24 hours
  A simple reaction time test which measures the participants' reaction time; they are looking at a red lamp, and need to react when it changes to green.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis B Zetner, MD, Principal Investigator — Center for Perioperative Optimization, Department of Surgery, Herlev Hospital, Denmark
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT03519750/Prot_SAP_000.pdf